CLINICAL TRIAL: NCT01355523
Title: The Effect of Melatonin on Depression, Anxiety, Cognitive Function and Sleep Disturbances in Breast Cancer Patients
Acronym: MELODY
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Inclusion rate not as expected. Not financially possible to involve other centres.
Sponsor: Melissa Voigt Hansen (Other)
Collaborators: University of Copenhagen (Other); Rigshospitalet, Denmark (Other); Pharma Nord (Industry)
Responsible Party: Sponsor-Investigator, Melissa Voigt Hansen, M.D., ph-D student, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MVH-03; 2010-022460-12 (EudraCT Number); 2007-58-0015/HEH.750.89-12 (Other: The Danish Data Protection Agency); H-4-2011-007 (Other: The Danish Ethics Committee)
Record Dates: First submitted 2011-05-13; First posted 2011-05-18 (Estimated); Results first posted 2014-05-06 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-04

CONDITIONS: Breast Cancer; Depression
Keywords: Breast cancer surgery; Melatonin; Depression; Anxiety; Sleep disturbances; Cognitive function
MeSH Terms: conditions — Breast Neoplasms; Depression; Anxiety Disorders; Parasomnias | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Melatonin (Active Comparator): 6 mg oral melatonin daily
  Interventions: Drug: Melatonin (N-acetyl-5-methoxytryptamine)
- Placebo (Placebo Comparator): 6 mg oral placebo daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Melatonin (N-acetyl-5-methoxytryptamine) — 6 mg oral melatonin daily 1 hour before bedtime
  Other Names: Melatonin; N-acetyl-5-methoxytryptamin
  Arms: Melatonin
Drug: Placebo — 6 mg oral placebo daily 1 hour before bedtime
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effect of 6 mg melatonin daily for 1 week preoperatively to 12 weeks postoperatively on depressive symptoms, anxiety, cognitive function and sleep disturbances in breast cancer patients. Furthermore the investigators will examine whether a specific clock-gene (HPER3) is correlated with an increased risk of depression, sleep disturbances or cognitive dysfunction.

DETAILED DESCRIPTION:
About 1.4 million women are diagnosed with breast cancer every year. Breast cancer is the most common malignancy among women worldwide constituting about 1/5 of all cancer types. Breast cancer diagnosis and treatment, and the months following primary therapy are stressful times for most women. Aside from the actual "cancer threat" many women experience various degrees of depression, anxiety, sleep disturbances and memory/concentration problems (cognitive dysfunction). Naturally these factors influence the quality of life but also contribute to morbidity and mortality.

Melatonin is a regulatory circadian hormone having, among others, hypnotic, sedative, anxiolytic and possibly anti-depressive effects. It has very low toxicity and very few adverse effects.

The purpose of this project is to test melatonin (6 mg daily for 1 week preoperatively to 12 weeks postoperatively) on breast cancer patients and hopefully hereby be able to prevent depression, anxiety, sleep disturbances and cognitive dysfunction. On an overall perspective this will hopefully contribute to improving the quality of life for these patients and extend their lifetime. Furthermore the investigators will be examining whether a specific gene called a clock-gene (HPER3) is correlated with an increased risk of depression, sleep disturbances or cognitive dysfunction. If this is the case it could become possible to identify women with an increased risk and provide prophylactic treatment for those with a risk of developing a depression, sleep disturbances or cognitive disturbances.

Sample size calculations were based on our primary outcome parameter. Using a conservative estimate for the incidence of depression, the investigators expect to find a reduction from 30% to 15% with melatonin treatment. Sample size is sufficient to include our secondary and tertiary outcome parameters as well. The sample size calculations were calculated with a power of 80%, a type I error of 5% and a type II error of 20%.

ELIGIBILITY:
Inclusion Criteria:

* Women, age 30-75, with breast cancer who are admitted for a lumpectomy or mastectomy at Herlev Hospital
* ASA score I-III
* No sign of depression measured my Major Depression Inventory (MDI)
* Not pregnant

Exclusion Criteria:

* Neoadjuvant chemotherapy
* Treatment with SSRI, Warfarin or other anticoagulants (except 75 mg ASA daily), MAO inhibitors or calcium blockers
* Rotor or Dubin-Johnson syndrome
* Epilepsy
* Known allergic reaction to melatonin
* Known and treated sleep apnea
* Diabetes Mellitus - insulin treated
* Ongoing or previous medically treated depression or bipolar disorder
* Known autoimmune diseases - systemic lupus erythematosus (SLE), rheumatoid arthritis (RA), and sclerose
* Incompensated liver cirrhosis
* Severe kidney disease
* Previous or current cancer
* Known medically treated sleep-disorder (insomnia, restless legs etc)
* Shift-work and night-work
* Daily alcohol intake of more than 5 units
* Pre-operative treatment with psychopharmacological drugs, opioids or anxiolytics (including all sleeping pills)
* Predicted bad compliance
* Pregnant or breast-feeding
* Pre-operative Mini Mental State Evaluation (MMSE) score less than 24

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2011-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa V Hansen, MD, Principal Investigator — Herlev Hospital
Locations (1):
- Herlev Hospital, Copenhagen, Denmark

REFERENCES:
- [Derived] Hansen MV, Madsen MT, Andersen LT, Hageman I, Rasmussen LS, Bokmand S, Rosenberg J, Gogenur I. Effect of Melatonin on Cognitive Function and Sleep in relation to Breast Cancer Surgery: A Randomized, Double-Blind, Placebo-Controlled Trial. Int J Breast Cancer. 2014;2014:416531. doi: 10.1155/2014/416531. Epub 2014 Aug 27. PMID 25328711

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was from July 2011 till December 2012. The location was The Department of Breast Surgery - Herlev Hospital, Copenhagen - Denmark.
Period: Overall Study
Arm/Group | Melatonin | Placebo
Started | 28 | 26
Completed | 27 | 16
Not Completed | 1 | 10
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Lost to Follow-up | 0 | 2
Not completed — Protocol Violation | 0 | 2
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Melatonin | Placebo | Total
Number analyzed (Participants) | 28 | 26 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 16 | 36
  >=65 years | 8 | 10 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.50 (10.69) | 58.23 (11.36) | 56.30 (11.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 26 | 54
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Denmark | 28 | 26 | 54
Type of surgery [Number; unit: Participants] — SN: sentinel node
  Participants
    Mastectomy + axillary dissection +/- SN | 1 | 3 | 4
    Mastectomy + SN | 4 | 3 | 7
    Lumpectomy + axillary dissection +/- SN | 6 | 6 | 12
    Lumpectomy + SN | 16 | 12 | 28
    Lumpectomy converted to mastectomy + SN | 1 | 0 | 1
    Bilateral lumpectomy + axillary dissection + SN | 0 | 2 | 2
Surgery duration [Median (Inter-Quartile Range); unit: Minutes] | 92 [74.5 to 125] | 125 [104.5 to 156.5] | 110 [85 to 141]
Anaesthesia duration [Median (Inter-Quartile Range); unit: Minutes] | 155 [130 to 187] | 190 [155 to 225] | 171 [139.25 to 196.25]
Oncological treatment [Number; unit: Participants] — Only registered as which oncological treatment (if any at all) the patients received during their participation in the MELODY trial
  Participants
    None | 3 | 3 | 6
    Radiation | 5 | 6 | 11
    Chemotherapy | 16 | 7 | 23
    Chemotherapy + radiation | 0 | 0 | 0
    Radiation x 1 only | 3 | 1 | 4
    Drop-out before chemo/radiation | 1 | 9 | 10
Anti-hormone therapy [Number; unit: Participants] — Only registered as which anti-hormone therapy (if any at all) the patients received during their participation in the MELODY trial
  Participants
    NO | 20 | 10 | 30
    YES | 7 | 7 | 14
    Drop-out before anti-hormone therapy | 1 | 9 | 10
MDI - Major Depression Inventory [Median (Inter-Quartile Range); unit: Scores on a scale] — The MDI is a self-rating scale including 12 questions and has been validated in a Danish population. The MDI assesses information on depressive symptoms that have been present continuously during the previous 2 weeks. The individual items are measured on a 6-point Likert scale, ranging from 0 to 5, with graduations depending on the extent of the symptom the previous 14 days. Accordingly, the theoretical score ranges from 0 to 50.
  Scores on a scale | 6.5 [4 to 12.5] | 7 [4.5 to 10] | 7 [4 to 11]
Menopausal status [Number; unit: Participants]
  Premenopausal | 14 | 10 | 24
  Postmenopausal | 14 | 16 | 30

OUTCOME MEASURES:

1. Primary Outcome: Major Depression Inventory (MDI)- Depression at One Point in the Study
Description: MDI is a self-rating depression scale with 12 questions. MDI has previously been investigated in a Danish population. On a six-point Likert scale, the items measure how much time the symptoms have been present during the last 14 days. MDI is scored according to specific guidelines and can be used either as a rating scale or diagnostic instrument.
  For inclusion we used the diagnostic instrument (depression was an exclusion criteria) and for all other MDI measurements we used the rating scale.
  Diagnostic scale using the ICD-10 algorithm:
  Mild depression: 2 core symptoms and 2 other symptoms Moderate depression: 2 core symptoms and 4 other symptoms Severe depression: 3 core symptoms and 5 other symptoms
  Rating scale:
  No depression - score from 0-20 Mild depression - score from 21-25 Moderate depression - score from 26-30 Severe depression - score from 31-50
Time Frame: Depression at one point in the study (not including baseline) out of 4 measurements at app. day 21, day 35, day 63 and day 91 of the study.
Population: Includes all patients who have completed at least one other MDI than baseline
Measure: Number; unit: participants
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 27 | 20
participants
  NO | 24 | 11
  YES | 3 | 9
Statistical Analysis 1: Comparison: Melatonin vs Placebo; Test type: Superiority or Other; p = 0.008, Chi-squared
Statistical Analysis 2: Comparison: Melatonin vs Placebo; Test type: Superiority or Other; Number need to treat = 2.95, 95% CI 2-sided [1.703 to 11.024]
Statistical Analysis 3: Comparison: Melatonin vs Placebo; Test type: Superiority or Other; Relative Risk = 0.25, 95% CI 2-sided [0.076 to 0.797]

2. Primary Outcome: Per Protocol - Depression at One Point in the Study Period
Description: MDI is a self-rating depression scale with 12 questions. MDI has previously been investigated in a Danish population. On a six-point Likert scale, the items measure how much time the symptoms have been present during the last 14 days. MDI is scored according to specific guidelines and can be used either as a rating scale or diagnostic instrument.
  For inclusion we used the diagnostic instrument (depression was an exclusion criteria) and for all other MDI measurements we used the rating scale.
  Rating scale:
  No depression - score from 0-20 Mild depression - score from 21-25 Moderate depression - score from 26-30 Severe depression - score from 31-50 This analysis includes only patients who have taken study medication as planned.
Time Frame: Per protocol - depression at one point in the study period (not baseline)
Population: Includes only patients who have taken the study medication as planned
Measure: Number; unit: participants
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 27 | 16
participants
  NO | 24 | 11
  YES | 3 | 5
Statistical Analysis 1: Comparison: Melatonin vs Placebo; Test type: Superiority or Other; p = 0.125, Fisher Exact

3. Primary Outcome: Intention to Treat (Underestimate) - Depression at One Point in the Study Period
Description: MDI is a self-rating depression scale with 12 questions. MDI has previously been investigated in a Danish population. On a six-point Likert scale, the items measure how much time the symptoms have been present during the last 14 days. MDI is scored according to specific guidelines and can be used either as a rating scale or diagnostic instrument.
  For inclusion we used the diagnostic instrument (depression was an exclusion criteria) and for all other MDI measurements we used the rating scale.
  Rating scale:
  No depression - score from 0-20 Mild depression - score from 21-25 Moderate depression - score from 26-30 Severe depression - score from 31-50 For this analysis all missing MDI data have been analyzed as "NO" depression.
Time Frame: Intention to treat (underestimate) - depression at one point in the study period (not baseline)
Population: All missing MDI data have been analyzed as "NO" depression.
Measure: Number; unit: participants
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 28 | 26
participants
  NO | 25 | 21
  YES | 3 | 5
Statistical Analysis 1: Comparison: Melatonin vs Placebo; Test type: Superiority or Other; p = 0.460, Fisher Exact

4. Primary Outcome: Intention to Treat (Overestimate) - Depression at One Point in the Study Period
Description: MDI is a self-rating depression scale with 12 questions. MDI has previously been investigated in a Danish population. On a six-point Likert scale, the items measure how much time the symptoms have been present during the last 14 days. MDI is scored according to specific guidelines and can be used either as a rating scale or diagnostic instrument.
  For inclusion we used the diagnostic instrument (depression was an exclusion criteria) and for all other MDI measurements we used the rating scale.
  Rating scale:
  No depression - score from 0-20 Mild depression - score from 21-25 Moderate depression - score from 26-30 Severe depression - score from 31-50 For this analysis all missing MDI data have been analyzed as "YES" for depression.
Time Frame: Intention to treat (overestimate) - depression at one point in the study period (not baseline)
Population: All missing data have been analyzed as "YES" depression.
Measure: Number; unit: participants
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 28 | 26
participants
  NO | 23 | 11
  YES | 5 | 15
Statistical Analysis 1: Comparison: Melatonin vs Placebo; Test type: Superiority or Other; p = 0.002, Chi-squared

5. Secondary Outcome: Area Under the Curve (AUC) for VAS Data on Anxiety - Immediate Postoperative Period
Description: Anxiety measured by VAS (visual analog scale). A subjective feeling of anxiety was registered on a VAS going from "no anxiety", equivalent to 0mm to "worst possible anxiety", equivalent to 100mm.
  Patients were only included in the analysis if they had completed daily VAS on anxiety, sleep quality, general well-being, fatigue, pain and sleepiness for at least 8 days postoperatively.
  Single missing data were filled out using last observation carried forward (LOCF). % of cases filled out by LOCF < 2 %
Time Frame: Daily - from inclusion till 8 days postoperatively
Measure: Median (Inter-Quartile Range); unit: mm*day
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 28 | 22
mm*day | 85 [44 to 160] | 140 [46 to 341]
Statistical Analysis 1: Comparison: Melatonin vs Placebo; Test type: Superiority or Other; p = 0.264, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Area Under the Curve (AUC) for VAS Data on Anxiety - Long-term Postoperative Period
Description: Anxiety measured by VAS (visual analog scale). Completed every 14th day. A subjective feeling of anxiety was registered on a VAS going from "no anxiety", equivalent to 0mm to "worst possible anxiety", equivalent to 100mm.
  Patients were only included in the analysis if they had completed VAS on anxiety, sleep quality, general well-being, fatigue, pain and sleepiness in the long-term postoperative period (every 14th day).
  Single missing data were filled out using last observation carried forward (LOCF). % of cases filled out by LOCF < 1 %
Time Frame: App. 14 days postoperatively till 10 weeks postoperatively
Population: Patients were only included in the analysis if they had completed VAS on anxiety in the long-term postoperative period. Single missing data were filled out using last observation carried forward.
Measure: Median (Inter-Quartile Range); unit: mm*2 weeks
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 27 | 16
mm*2 weeks | 14 [4 to 31] | 19 [8 to 100]
Statistical Analysis 1: Comparison: Melatonin vs Placebo; Test type: Superiority or Other; p = 0.351, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Area Under the Curve (AUC) for Data on Sleepiness (KSS) - Immediate Postoperative Period
Description: Sleepiness measured by Karolinska Sleepiness Scale. KSS is a 9-point scale from 1 (very awake) to 9 (very sleepy) where a score of 7 or more reflects pathological sleepiness.
  Patients were only included in the analysis if they had completed daily VAS on anxiety, sleep quality, general well-being, fatigue, pain and sleepiness for at least 8 days postoperatively.
  Single missing data were filled out using last observation carried forward (LOCF). % of cases filled out by LOCF < 2 %
Time Frame: Daily from inclusion till 8 days postoperatively
Measure: Median (Inter-Quartile Range); unit: Units on KSS*day
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 28 | 22
Units on KSS*day | 35 [26 to 48] | 39 [31 to 55]
Statistical Analysis 1: Comparison: Melatonin vs Placebo; Test type: Superiority or Other; p = 0.446, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Area Under the Curve (AUC) for Data on Sleepiness (KSS) - Long-term Postoperative Period
Description: Sleepiness measured by Karolinska Sleepiness Scale. KSS is a 9-point scale from 1 (very awake) to 9 (very sleepy) where a score of 7 or more reflects pathological sleepiness.
  Patients were only included in the analysis if they had completed VAS on anxiety, sleep quality, general well-being, fatigue, pain and sleepiness in the long-term postoperative period (every 14th day).
  Single missing data were filled out using last observation carried forward (LOCF). % of cases filled out by LOCF < 1 %
Time Frame: App. 14 days postoperatively till 10 weeks postoperatively
Measure: Median (Inter-Quartile Range); unit: Units on KSS*2 weeks
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 27 | 16
Units on KSS*2 weeks | 13 [11 to 17] | 14 [12 to 20]
Statistical Analysis 1: Comparison: Melatonin vs Placebo; Test type: Superiority or Other; p = 0.122, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Area Under the Curve (AUC) for VAS Data on Fatigue - Immediate Postoperative Period
Description: Fatigue on a Visual Analog Scale - filled out daily. A subjective feeling of fatigue was registered on a VAS going from "no fatigue", equivalent to 0mm to "worst possible fatigue", equivalent to 100mm.
  Patients were only included in the analysis if they had completed daily VAS on anxiety, sleep quality, general well-being, fatigue, pain and sleepiness for at least 8 days postoperatively.
  Single missing data were filled out using last observation carried forward (LOCF). % of cases filled out by LOCF < 2 %
Time Frame: Daily from inclusion till 8 days postoperatively
Measure: Median (Inter-Quartile Range); unit: mm*day
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 28 | 22
mm*day | 307 [93 to 399] | 300 [146 to 429]
Statistical Analysis 1: Comparison: Melatonin vs Placebo; Test type: Superiority or Other; p = 0.907, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Area Under the Curve (AUC) for VAS Data on Fatigue - Long-term Postoperative Period
Description: Fatigue on a Visual Analog Scale - filled out every 14th day. A subjective feeling of fatigue was registered on a VAS going from "no fatigue", equivalent to 0mm to "worst possible fatigue", equivalent to 100mm.
  Patients were only included in the analysis if they had completed VAS on anxiety, sleep quality, general well-being, fatigue, pain and sleepiness in the long-term postoperative period (every 14th day).
  Single missing data were filled out using last observation carried forward (LOCF). % of cases filled out by LOCF < 1 %
Time Frame: App. 14 days postoperatively till 10 weeks postoperatively
Measure: Median (Inter-Quartile Range); unit: mm*2 weeks
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 27 | 16
mm*2 weeks | 90 [58 to 147] | 88 [41 to 133]
Statistical Analysis 1: Comparison: Melatonin vs Placebo; Test type: Superiority or Other; p = 0.555, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Area Under the Curve (AUC) for Data on General Well-being - Immediate Postoperative Period
Description: General well-being on a Visual Analog Scale - filled out daily. A subjective feeling of general well-being was registered on a VAS going from "very high well-being", equivalent to 0mm to "very low well-being", equivalent to 100mm.
  Patients were only included in the analysis if they had completed daily VAS on anxiety, sleep quality, general well-being, fatigue, pain and sleepiness for at least 8 days postoperatively.
  Single missing data were filled out using last observation carried forward (LOCF). % of cases filled out by LOCF < 2 %
Time Frame: Daily from inclusion till 8 days postoperatively
Population: Patients were only included in the analysis if they had completed daily VAS on anxiety for at least 8 days postoperatively. Single missing data were filled out using last observation carried forward.
Measure: Median (Inter-Quartile Range); unit: mm*day
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 28 | 22
mm*day | 282 [211 to 436] | 372 [180 to 450]
Statistical Analysis 1: Comparison: Melatonin vs Placebo; Test type: Superiority or Other; p = 0.930, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Area Under the Curve (AUC) for VAS Data on General Well-being - Long-term Postoperative Period
Description: General well-being on a Visual Analog Scale - filled out every 14th day. A subjective feeling of general well-being was registered on a VAS going from "very high well-being", equivalent to 0mm to "very low well-being", equivalent to 100mm.
  Patients were only included in the analysis if they had completed VAS on anxiety, sleep quality, general well-being, fatigue, pain and sleepiness in the long-term postoperative period (every 14th day).
  Single missing data were filled out using last observation carried forward (LOCF). % of cases filled out by LOCF < 1 %
Time Frame: App. 14 days postoperatively till 10 weeks postoperatively
Measure: Median (Inter-Quartile Range); unit: mm*2 weeks
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 27 | 16
mm*2 weeks | 95 (141) [52 to 141] | 89 (44) [44 to 142]
Statistical Analysis 1: Comparison: Melatonin vs Placebo; Test type: Superiority or Other; p = 0.386, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Area Under the Curve (AUC) for VAS Data on Pain - Immediate Postoperative Period
Description: Pain on a Visual Analog Scale - filled out daily. A subjective feeling of pain was registered on a VAS going from "no pain", equivalent to 0mm to "worst possible pain", equivalent to 100mm.
  Patients were only included in the analysis if they had completed daily VAS on anxiety, sleep quality, general well-being, fatigue, pain and sleepiness for at least 8 days postoperatively.
  Single missing data were filled out using last observation carried forward (LOCF). % of cases filled out by LOCF < 2 %
Time Frame: Daily from inclusion till 8 days postoperatively
Measure: Median (Inter-Quartile Range); unit: mm*day
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 28 | 22
mm*day | 97 [45 to 181] | 130 [46 to 421]
Statistical Analysis 1: Comparison: Melatonin vs Placebo; Test type: Superiority or Other; p = 0.241, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Area Under the Curve (AUC) for VAS Data on Pain - Long-term Postoperative Period
Description: Pain on a Visual Analog Scale - filled out every 14th day. A subjective feeling of pain was registered on a VAS going from "no pain", equivalent to 0mm to "worst possible pain", equivalent to 100mm.
  Patients were only included in the analysis if they had completed VAS on anxiety, sleep quality, general well-being, fatigue, pain and sleepiness in the long-term postoperative period (every 14th day).
  Single missing data were filled out using last observation carried forward (LOCF). % of cases filled out by LOCF < 1 %
Time Frame: App. 14 days postoperatively till 10 weeks postoperatively
Measure: Median (Inter-Quartile Range); unit: mm*2 weeks
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 27 | 16
mm*2 weeks | 13 [2 to 48] | 22 [8 to 76]
Statistical Analysis 1: Comparison: Melatonin vs Placebo; Test type: Superiority or Other; p = 0.339, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Area Under the Curve (AUC) for VAS Data on Sleep Quality - Immediate Postoperative Period
Description: Subjective sleep score on Visual Analog Scale. Subjective sleep quality was registered on a VAS going from "best possible sleep", equivalent to 0mm to "worst possible sleep", equivalent to 100mm.
  Patients were only included in the analysis if they had completed daily VAS on anxiety, sleep quality, general well-being, fatigue, pain and sleepiness for at least 8 days postoperatively.
  Single missing data were filled out using last observation carried forward (LOCF). % of cases filled out by LOCF < 2 %
Time Frame: Daily from inclusion till 8 days postoperatively
Measure: Median (Inter-Quartile Range); unit: mm*day
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 28 | 22
mm*day | 279 [203 to 466] | 355 [194 to 441]
Statistical Analysis 1: Comparison: Melatonin vs Placebo; Test type: Superiority or Other; p = 0.578, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Area Under the Curve (AUC) for VAS Data on Sleep Quality - Long-term Postoperative Period
Description: Subjective sleep on a Visual Analog Scale. Subjective sleep quality was registered on a VAS going from "best possible sleep", equivalent to 0mm to "worst possible sleep", equivalent to 100mm.
  Patients were only included in the analysis if they had completed VAS on anxiety, sleep quality, general well-being, fatigue, pain and sleepiness in the long-term postoperative period (every 14th day).
  Single missing data were filled out using last observation carried forward (LOCF). % of cases filled out by LOCF < 1 %
Time Frame: App. 14 days postoperatively till 10 weeks postoperatively
Measure: Median (Inter-Quartile Range); unit: mm*2 weeks
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 27 | 16
mm*2 weeks | 101 [51 to 148] | 116 [51 to 133]
Statistical Analysis 1: Comparison: Melatonin vs Placebo; Test type: Superiority or Other; p = 1.000, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: Sleep Architecture
Description: Actigraphy (total minutes asleep, sleep effectiveness, sleep latency, awakenings). A wrist actigraph will be worn from inclusion till 14 days postoperatively.
Time Frame: From inclusion till 14 days postoperatively
Reporting Status: Not Posted

18. Secondary Outcome: HPER3 Genotype
Description: A blood sample will be taken at inclusion and analysed for HPER3 genotype (4/4, 4/5, 5/5) and this will be investigated for a correlation with sleep, cognitive function and depressive symptoms 7 patients did not give blood samples
Time Frame: At inclusion = day-7
Measure: Number; unit: Participants
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 26 | 21
Participants
  4/4 genotype | 14 | 10
  4/5 genotype | 10 | 10
  5/5 genotype | 2 | 1
  Missing | 2 | 5

19. Secondary Outcome: Incidence of Postoperative Cognitive Dysfunction (POCD) App. 2 Weeks Postoperatively.
Description: Calculations for POCD were based on normative data from 133 females aged 40-60 years. We evaluated changes from the preoperative baseline to the 2 postoperative test sessions. In controls we calculated mean and standard deviations (SD) of these differences. The mean change in this group may be taken as estimated learning effects. For the individual patients, we compared baseline scores with the 2- and 12-week postoperative test results, subtracted the average learning effect from the changes and divided the result by the SD of the control group to obtain a Z score for the 7 individual test outcomes. A large positive Z score indicated deterioration in cognitive function from baseline in patients. We defined a composite Z score as the sum of the 7 Z scores and normalized this using the SD for that sum in the controls. POCD was defined as a combined Z score >1.96 or a Z score >1.96 in at least 2 of the 7 subtests.
  Units of measure = % of patients with YES to POCD
Time Frame: App. 2 weeks postoperatively
Population: Analysis includes only patients who completed all parts of the neuropsychological test battery at baseline and 2 weeks postoperatively.
Measure: Number; unit: Percentage of patients
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 26 | 20
Percentage of patients | 0 | 0

20. Secondary Outcome: Incidence of Postoperative Cognitive Dysfunction (POCD) App. 10 Weeks Postoperatively
Description: as for outcome 19
Time Frame: App. 10 weeks postoperatively
Population: Analysis includes only patients who completed all parts of the neuropsychological test battery at baseline and 10 weeks postoperatively.
Measure: Number; unit: Percentage of patients
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 26 | 16
Percentage of patients | 0 | 6.25

ADVERSE EVENTS:
Time Frame: From inclusion (app. 1 week preoperatively) till the final visit (app. 10 weeks postoperatively)
Description: Only includes patients who have at least taken 1 dose of the study drug.
Arm/Group | Melatonin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/24
Other Adverse Events (participants affected / at risk) | 15/27 | 9/24
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Melatonin (N=27) | Placebo (N=24)
Headache (Nervous system disorders) | 3 | 4
Dizziness (Ear and labyrinth disorders) | 4 | 1
Sleepiness (Nervous system disorders) | 1 | 1
Difficulty falling asleep (General disorders) | 1 | 2
More awakenings at night (General disorders) | 1 | 0
Tiredness (General disorders) | 1 | 0
Paraesthesia (mouth region, arms/legs) (Nervous system disorders) | 3 | 0
Memory problems (Nervous system disorders) | 1 | 0
Breathing difficulties (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2
Reflux (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Dry mouth (Skin and subcutaneous tissue disorders) | 1 | 0
Obstipation (Gastrointestinal disorders) | 1 | 0
Vomitus (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Urinary urgency (Renal and urinary disorders) | 1 | 0
Diffuse pain in the lower abdomen (Gastrointestinal disorders) | 1 | 0
Lower back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Flushing/sweating (Skin and subcutaneous tissue disorders) | 2 | 1
Itch (arms) (Musculoskeletal and connective tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Premature termination (54/260). Only included about 8% (54/703) of the patients assessed for eligibility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No